CLINICAL TRIAL: NCT07006259
Title: Effect of Bobath Therapy on Balance Alterations in Patients With Multiple Sclerosis
Acronym: BTPCMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Neurofis
Record Dates: First submitted 2025-05-07; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Bobath Therapy; Postural Control; Virtual Reality; Home Exercise Program

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): Treatment with bobath Therapy
  Interventions: Other: Bobath Therapy
- Experimental group A (Active Comparator): Bobath Therapy plus Virtual Reality
  Interventions: Other: Bobath therapy plus virtual reality
- Experimental group B (Active Comparator): Home exercises
  Interventions: Other: Home exercises

INTERVENTIONS:
Other: Bobath Therapy — Treatment with bobath therapy
  Arms: Control group
Other: Bobath therapy plus virtual reality — Treatment with bobath therapy plus virtual reality
  Arms: Experimental group A
Other: Home exercises — Treatment with home exercises
  Arms: Experimental group B

SUMMARY:
To evaluate the effects of a foot treatment to improve balance according to the Bobath Concept in people with Multiple sclerosis, comparing it with treatment through home exercise and with treatment from Bobath Concept combined with the use of virtual reality.

As a secondary objective, we seek to know the state of the art of Bobath therapy in Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age: over 18 years old.
2. Have a diagnosis of multiple sclerosis, according to Mc Donald criteria at least 6 months before the start of the intervention.
3. Be able to walk independently in a closed environment with or without technical aids, having a maximum score of 6.5 on the Expanded Disability Status Scale or EDSS, according to its acronym in English:

6.5= constant bilateral help (canes, crutches or braces) to walk about 20 meters without rest. The usual functional system (FS) is equivalent to combinations with more than two FS of grade 3+.

Exclusion Criteria:

1. Participants who are not able to understand instructions,
2. Participants who are in a clinically unstable situation or who have risk factors or concomitant pathologies of the musculoskeletal system, neurological or cardiovascular, which make it difficult to carry out the treatment.
3. Participants with visual disturbances or severe upper limb involvement who therefore have difficulty using the VR glasses or performing reaching exercises with them.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Balance Evaluation Systems Test (Mini BESTest). | At the beginning, at the month and we would reevaluate after 15 days
  It assesses balance in six items (biomechanical restrictions, stability and verticality limits, anticipatory postural adjustments, postural responses, sensory orientation, and gait stability). It has excellent inter- and intra-observer reliability and construct validity in stroke patients. Furthermore, the items on anticipatory postural adjustments and sensory orientation are highly correlated with the risk of falls in this type of pathology.

SECONDARY OUTCOMES:
Timed Up and Go Test | At the beginning, at the month and we would reevaluate after 15 days
  It assesses the risk of falls. It allows the measurement of functional movement. It has excellent inter- and intra-observer reliability and good construct validity. A test duration of more than 13.5 seconds is associated with an elevated risk of falls

OTHER OUTCOMES:
Functional reach test (FRT) | At the beginning, at the month and we would reevaluate after 15 days
  It is one of the most widely used balance scales because it measures the limits of stability in standing. It also identifies limitations in activities of daily living (ADLs) and indicates the risk of falls. The final FRT score is the distance between the initial and final positions. Results of less than 25 cm indicate a limitation in ADLs and a risk of falls.
Modified Fatigue Impact Scale (MFIS) | At the beginning, at the month and we would reevaluate after 15 days
  The MFIS uses a multidimensional approach with cognitive, physical, and psychosocial components. It consists of approximately 21 items in the form of questions related to the patient's feeling of fatigue. The maximum possible score is 84, with higher scores indicating a greater impact on quality of life.
MusiQoL | At the beginning, at the month and we would reevaluate after 15 days
  The Spanish version of the MusiQoL questionnaire appears to be a valid and reliable instrument for measuring quality of life in MS patients in Spain and is a useful tool for measuring health-related quality of life in the clinical setting. The MusiQoL is a questionnaire used to assess quality of life in people with multiple sclerosis. To score, the responses to the items are added together to obtain a total score, which can range from 0 to 100. The higher the score, the higher the perception of quality of life.
Neo-plate pressure platform | At the beginning, at the month and we would reevaluate after 15 days
  A static analysis of pressure distribution will be performed with the patient standing, differentiating between forefoot and hindfoot loads, and between the right and left feet, as well as by quadrant, and quantifying the deviation from the center of pressure position. A dynamic analysis will be performed during gait, recording contact time, average pressure, and the time/contact integral. Several studies demonstrate the use of pedometric platforms to assess and improve gait and balance disorders in patients with MS. The Neo-plate pressure platform can measure mean and maximum pressures in kPa, stabilometry and oscillation data of the center of pressure in mm/s and the force exerted by the foot during walking in kg.
Computerized dynamic posturography (PDC). | At the beginning, at the month and we would reevaluate after 15 days
  It is a quantitative method for the assessment and treatment of balance disorders. It is based on the use of dynamometric platforms that measure the displacement of the center of pressure by collecting the sensors located on it, the different pressure stimuli exerted by the subject's body in different static and dynamic situations and is considered by several authors as the gold standard for the study of postural control.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided